CLINICAL TRIAL: NCT00509704
Title: Pilot Study on the Influence of Sutent on Tumor Vascularization and Necrosis in Patients With Renal Cell Carcinoma
Brief Title: Influence of Sutent on Tumor Vascularization and Necrosis in Patients With Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: C.M.L. van Herpen,, University Medical Centre Nijmegen, st Radboud
Other Study IDs: CMO 2006/232
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-10

CONDITIONS: Renal Cell Cancer
Keywords: Sutent; tumor necrosis; DCE-MRI (Dynamic enhanced magnetic resonance imaging)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to assess the effect of Sunitinib on tumor vascularization and necrosis in patients with metastatic renal cell cancer.

DETAILED DESCRIPTION:
Sutent is an angiogenesis inhibitor used in the treatment of renal cell cancer. Very often tumor necrosis is seen after the start of the treatment. It is unknown after how many days this effect starts. In patients with renal cell cancer with metastases, who will be treated with Sutent, 3 MRIs will be made. Kep, R2*, b-coefficient (perfusion, hypoxia, blood volume and necrosis) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* patients with metastatic renal cell cancer for whom treatment with Sunitinib is planned
* histologically verified stage IV renal cell carcinoma of clear cell type
* measurable primary tumor or metastases (minimal diameter 2 cm) at other sites than the lungs
* Karnofsky score > 70%
* age > 18 year.
* written informed consent

Exclusion Criteria:

* contra-indications for MRI
* contra-indications for treatment with Sunitinib
* previous systemic treatment within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a malignant abdominal tumor or metastases (minimal diameter 2 cm)
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2008-10; Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, MD, PhD, Principal Investigator — UMC St Radboud
Locations (1):
- UMC St Radboud, Nijmegen, Netherlands